CLINICAL TRIAL: NCT05904821
Title: Relationship Between BMI, Physical Fitness and Motor Skills in Children With Down's Syndrome
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC/RCR & AHS/23/0706
Record Dates: First submitted 2023-06-06; First posted 2023-06-15 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Down Syndrome
Keywords: BMI; Down Syndrome; Motor Skills; Physical Fitness; Test of Gross Motor Development (TGMD-2); SAMU Disability Fitness Battery (SAMU-DISFIT)
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Down syndrome is a congenital condition which includes physical mental, and functional abnormalities. It arises from defect involving chromosome 21, usually an extra copy (trisomy 21). Purpose of this study will determine the relationship between BMI, physical fitness and motor skills in youth with down syndrome

DETAILED DESCRIPTION:
This will be a cross-sectional study. The sample size is 169. The inclusion criteria will be Diagnosed with trisomy 21, Aged 6-11 years, Abel to follow a minimum of two-step instructions, The minimum motor ability of participants with DS is independent locomotion where as the exclusion criteria will be medical condition that is contraindicated to moderate to vigorous physical activity such as cardiovascular problems, orthopedic instability, including those associated with DS (e.g., Atlanto-axial instability), behavioral issues that hindered instruction. The BMI will be assessed using a person's height and weight. The formula is BMI = kg/m 2 where kg is a person's weight in kilograms and m 2 is their height in meters squared. Physical Fitness by using SAMU Disability Fitness Battery (SAMU-DISFIT). the Timed Up and Go test (TUG), the Deep Trunk Flexibility test (DTF), the Hand Grip test (HG), the Timed Stand Test (TST), the 30-s Sit-Up (SUP), the 6-Min Walk Test (6MWT) and Motor Skills using Test of Gross Motor Development (TUG-2) Data will be analyzed using SPSS 22.0. Frequency tables and bar charts will be used for descriptive statistics Chi-Square will be used to find the Association

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with trisomy 21.
* Aged 5-15 years.
* Abel to follow a minimum of two-step instructions.
* The minimum motor ability of participants with DS is independent locomotion.

Exclusion Criteria:

* Medical condition that is contraindicated to moderate to vigorous physical activity such as cardiovascular problems.
* Orthopedic instability, including those associated with DS (e.g., Atlanto-axial instability).
* Behavioral issues that hindered instruction

Ages: 4 Years to 15 Years | Sex: All
Age Groups: Child
Study Population: DownsSyndrome
Sampling Method: Non-Probability Sample
Enrollment: 169 (Actual)
Dates: Start 2023-05-23 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Time up and go (TUG) | 2 months
  The participant will sit in a chair keeping the back straight in contact with the backrest, the feet resting on the floor and the hands on the thighs. At the "go" signal, the subject gets up from the chair, moves as fast as he can to the line fifteen black that is located 3 m from the front legs of the chair, turns and returns to the sitting position traveling a total of 6 m (3 out and 3 back). The timer starts when the subject starts to move and stops when the back touches the back when sitting down.
The Deep Trunk Flexibility test (DTF) | 2 months
  The initial position of the subjects was standing with their legs separated at the width of the waist. The subjects flexed their trunk and their knees and put their arms downwards and behind their legs to slide the cursor of the millimeter bar with their fingertips of both hands. A measurement bench (10 × 10 × 55 cm, height, width and length, respectively) was used for the evaluation. Two tries were done, and the best mark was chosen, following the indications of Valdivia et al. with children and adolescents
The Hand Grip test (HG). | 2 months
  The subject is placed in a standing position with the dynamometer in his dominant hand. The dynamometer grip is adjusted to the size of the hand to have the second phalanx of the index finger approximately at a right angle. Arms slightly separated from the body. It is not allowed to lean the trunk to any side or bend the elbows. The subject squeezes the dynamometer firmly and gradually, rapidly increasing to maximum force muscles, especially of the finger flexors. The participants were asked to push as hard as possible after the command 'and go'. There were two tries with each hand, establishing 10 s of rest between them
Timed Stand Test (TST). | 2 months
  The subject must sit on the chair so that his knees form an angle of 90º. To do this, it will be necessary to adjust the height of the chair for each participant. The subject sits in the chair, which will be leaning against a wall, and is asked to perform ten squats as quickly as possible without using the arms to propel himself. The arms should remain crossed in front of the chest and straighten the knees with each repetition. The timer starts when the movement is started and stops when the subject returns to a sitting position after the tenth squat. Rubber treads may be used to facilitate foot placement for the subject
The 30-s Sit-Up (SUP). | 2 months
  The subject must be lying in a supine position with the legs resting on the floor.
  The maximum number of push-ups should be performed for 30 seconds. The correct execution (what is considered a correct complete repetition) is established when the participant raises the scapulae from the ground, keeping the arms stretched out in front and resting them again. As a reference, it was indicated that the subjects touch the patella (put the evaluator's arm in that area to avoid confusion), which in this position forces the scapular area to come off the ground. It is recommended that the investigator hold the participant's legs to prevent any movement of her legs or feet
The 6-Min Walk Test (6MWT) | 2 months
  : Regarding the use of the clock, follow the manufacturer's instructions for its correct operation. The participant must try to cover the maximum distance possible in 6 minutes. Running is prohibited, so the subject can only walk fast. It is necessary that the research staff constantly motivate the participants
BMI (BMI = kg/m2) | 2 months
  To calculate the BMI, the weight (kg) is divided by the height (m2) difference is greater than 1cm/1kg, a third measurement will be taken. Subsequently, the average is made with the two closest measurements.
Waist Circumference | 2 months
  The subject will be standing, with the abdomen relaxed and the arms relaxed parallel to the trunk. The measurement should not be done on clothing, so the shirt should be removed or pulled up without you having to hold it. From this position, the examiner will encircle the subject's waist with the tape measure. The measurement will be made at the narrowest level, between the edge of the lower costal (10th rib) and the iliac crest, at the end of a normal expiration and without the tape pressing on the skin and with the participant's arms at their sides. If there is no obvious minimum waist, the measurement will be taken at the midpoint between the lower costal edge (10th rib) and the iliac crest.
ROM | 2 months
  The subject will be placed in a standing position with the legs separated at the width of the hips. The feet will be in line with the edge of the instrument, so that the heels are placed on the line at the 0 level of the scale, and they will not be able to move during the test. At the signal, the person must flex the trunk downwards and backwards, pushing the cursor of the millimeter bar with the middle fingers of both hands (which have passed between the legs) until they advance as far as possible. It is allowed to flex the knees
Run | 2 months
  Directions:Mark off two lines 50 feet apart. Instruct student to "run fast" from one line to the other.
  "Brief period where both feet are off the ground "Arms in opposition to legs, elbows bent. Foot placement near or on line (not flat footed). onsupport leg bent approximately 90 degrees (close to buttocks).
Gallop | 2 months
  Mark off two lines 30 feet apart. Tell student to gallop from one line to the other three times. Tell student to gallop leading with one foot and then the other. A step forward with the lead foot followed by a step with the trailing foot to a position adjacent to or behind the led foot.
  * "Brief period where both feet are off the ground.
  * "Arms bent and lifted to waist level.
Hop | 2 months
  DIRECTIONS: Ask the student to hop three times, first on one foot and then on the other.
  *This criteria does not require the performance of the other three. Foot of nonsupport leg is bent and carried in back of the body.
  * "Nonsupport leg swings in pendular fashion to produce force.
  * "Arms bent at elbows and swing forward on take off.
  * "Able to hop on the right and left foot.*
Leap | 2 months
  DIRECTIONS: Ask the student to leap. Tell the student to take large steps by leaping from one foot to the other.
  Take off on one foot and land on the opposite foot.
  * "A period where both feet are off the ground (longer than running).
  * "Forward reach with arm opposite the lead foot.
Horizontal Jump | 2 months
  DIRECTIONS: Mark off a starting line on the floor, mat, or carpet. Have the student start behind the line. Tell the student to "jump far."
  * "Preparatory movement includes flexion of both knees with arms extended behind the body.
  * "Arms extend forcefully forward and upward, reaching full extension above head.
  * "Take off and land on both feet simultaneously.
  * "Arms are brought downward during landing.
Skip | 2 months
  DIRECTIONS: Mark off two lines 30 feet apart. Tell the student to skip from one line to the other three times.
  * "A rhythmical repetition of the step-hop on alternate feet.
  * "Foot of nonsupport leg carried near surface during hop phase.
  * "Arms alternately moving in opposition to legs at about waist level
Slide | 2 months
  DIRECTIONS: Mark off two lines 30 feet apart. Tell the student to slide from one line to the other line three times facing the same direction.
  "Body turned sideways to desired direction of travel.
  * "A step sideways followed by a slide of the trailing foot to a point next to the lead foot.
  * "A short period where both feet are off the floor.
  * "Able to slide to the right and to the left side.
Two Hand strike | 2 months
  DIRECTIONS: Toss the ball softly to the student at bout waist level. Tell the student to hit the ball"hard." Count only those tosses that are between the student's waist and shoulders.
  * "Dominant hand grips bat above nondominant hand.
  * "Nondominant side of body faces the tosser (feet parallel).
  * "Hip and spine rotation.
  * "Weight is transferred by stepping with front foot.
Stationary Bounce | 2 months
  DIRECTIONS: Tell the student to bounce the ball three times using one hand. Make sure the ball is not underinflated. Repeat three separate trials.
  * "Contact ball with one hand at about hip height.
  * "Pushes ball with fingers (not a slap).
  * "Ball contacts floor in front of (or to the outside of) foot on the side of the hand being used.
Catch | 2 months
  DIRECTIONS: Mark off two lines 15 feet apart. Student stands on one line and the tosser on the other. Toss the ball underhand directly to student with a slight arc, saying "catch it with your hands." Only count those tosses that are between student's shoulders and waist.
  "Preparation phase where elbows are flexed and hands are in front of body.
  * "Arms extend in preparation for ball contact.
  * "Ball is caught and controlled by hands only.
  * "Elbows bend to absorb force
kick | 2 months
  DIRECTIONS: Mark off one line 30 feet away from a wall and one that is 20 feet from the wall. Place the ball on the line nearest the wall and tell the student to stand on the other line. Tell the student to kick the ball "hard" toward the wall.
  * "Rapid continuous approach to the ball.
  * "The trunk is inclined backward during ball contact.
  * "Forward swing of the arm opposite kicking leg.
  * "Follow-through by hopping on non-kicking foot.
Overhead Throw | 2 months
  DIRECTIONS: Tell the student to throw the ball "hard" at the wall.
  * "A downward arc of the throwing arm initiates the windup.
  * "Rotation of hip and shoulder to a point where the nondominant side faces an imaginary target.
  * "Weight is transferred by stepping with the foot
  * "Follow-through beyond ball release diagonally across body toward side opposite throwing arm.

CONTACTS AND LOCATIONS:
Overall Officials: Mahnoor Bukhari, MS, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No